CLINICAL TRIAL: NCT06345573
Title: Sex Differences in Heart-brain Crosstalk - Role of Psychosocial Stress
Brief Title: Heart-brain-axis and Psychosocial Stress
Status: Active, not recruiting | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2020-02922
Record Dates: First submitted 2024-03-05; First posted 2024-04-03 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Mental Stress; Myocardial Ischemia; Sex Role; Gender
MeSH Terms: conditions — Stress, Psychological; Myocardial Ischemia; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female Sex: Healthy volunteer women aged between 50-75 years old, in post-menopausal status.
  Interventions: Behavioral: Mental stress
- Male Sex: Healthy volunteer men aged between 50-75 years old.
  Interventions: Behavioral: Mental stress

INTERVENTIONS:
Behavioral: Mental stress — Two consecutive validated mental stress tests, namely 1) the Montreal Imaging Stress Task consisting of two series of 15-minute mental calculation tests, without (Control Mode) and with (Stress Mode) negative feedback, respectively; and 2) the Trier Social Stress Test consisting of a 5-minute mock job interview (Speech Part) followed by a 5-minute mental calculation test (Mental Arithmetic Part).

SUMMARY:
The main study objective is to prospectively determine the influence of sex-related risk factors and psychosocial variables on neuronal stress responses and myocardial perfusion in a population of 64 female and male individuals 50-75 years of age and free of cardiovascular disease.

DETAILED DESCRIPTION:
The main objective of the project is to prospectively determine the influence of sex on amygdalar metabolic activity and myocardial perfusion in a population of healthy postmenopausal women and aged men under acute psychosocial stress conditions.

The primary hypothesis of the study is that women experience disproportionate amygdalar metabolic activity and reduced myocardial perfusion in response to psychosocial stress compared to men.

This project is a monocentric prospective observational study involving hybrid positron emission tomography/magnetic resonance (PET/MR) imaging as well as the collection of biological samples in healthy individuals aged 50-75 years (postmenopausal women, and men). To inflict acute psychosocial stress, the investigators applied the Montreal Imaging Stress Test (MIST) when the participants were inside the PET/MR scanner and the Trier Social Stress Test (TSST) when the participants were outside the PET/MR scanner. Both the TSST and the MIST are standardized tests and are widely applied to provoke reliable biological stress responses in a laboratory setting. No follow-up study is planned. At inclusion, individuals have been interviewed and health data have been collected through questionnaires. In addition, biological samples, including blood, nail and saliva have been collected. Volunteers underwent myocardial blood flow (MBF) and cerebral perfusion imaging using ammonia (13NH3)-PET, as well as functional imaging using magnetic resonance imaging (MRI), both routinely used imaging techniques. 13NH3-PET/MR has been conducted at rest and under stress (MIST). Subsequently, the study participants underwent a TSST, followed by whole body metabolic imaging with fluor-18-deoxyglucose (18F-FDG)-PET/MRI, allowing to study brain and bone marrow metabolism, among other parameters. In parallel, the heart rate response (HRR) has been monitored throughout the study and catecholamines were collected at baseline and after stress to assess the autonomic influence on the heart. The total radiation exposure was below 5 mSv.

In detail, each participant was asked to complete questionnaires to assess their psychometric baseline characteristics at the study visit.

Two blood samples were collected from a peripheral intravenous catheter, at the beginning of the study and the end of the TSST. Blood glucose levels were measured using a finger prick. In addition, saliva samples of approximately 1 mL each were taken at different time points, notably before and after each of the mental stress tests. Nail samples were collected by clipping nails from the fingers and/or toes.

All biological samples from the participants were immediately processed to allow sample conservation.

Project data and samples were handled with the uttermost discretion and only accessible to authorized personnel. On project-specific documents, participants are only identified by a unique participant number. Coded data were used and the participant identification list is only accessible by the investigators. Data is protected from unauthorized or accidental disclosure, alteration, deletion, copying, and theft by using the built-in mechanisms of Redcap®. Biological material in this project is not identified by participant name but by a unique participant number.

Participants were asked to fast for at least 2.5 hours prior to the study visit and refrain from strong physical activity for at least 24 hours. All study participants underwent serial imaging on a dedicated hybrid PET/MR scanner (GE Healthcare) using 13N-NH3 and 18F-FDG as validated tracers, according to daily clinical routine. Whole-body (18F-FDG) or brain and heart (13-NH3) MRI were recorded simultaneously with all PET scan acquisitions. Beginning with an intravenous bolus administration of 200 MBq of 13N-NH3, serial dynamic and static PET images were acquired for 30 minutes. In parallel, subjects underwent the Control (rest) part of the MIST (mathematical task, inside the scanner). A second dose of 400 MBq of 13N-NH3 was given, and images were recorded in the same acquisition sequence for 30 minutes, in parallel to the Stress part of the MIST.

After a break, all individuals were injected with 150 MBq of 18F-FDG, followed by a TSST outside of the scanner. During the first part of the TSST, a panel of two to three judges (trained staff), equipped with a video camera, ask the participant to prepare a 5-minute presentation. To do that, participants can use paper and pen but must hand out their notices at the beginning of the presentation. During the 5-minute presentation, the judges observe the participants without giving any comments or facial expressions. The participants are asked to continue if they stop before the entire 5 minutes run out. For the second part of the TSST, participants undergo a mental arithmetic task during which they are asked to count backward from 1022 in steps of 11. Subsequently, participants were allowed to rest in a designated separate dark room (rest phase), and the 18F-FDG-PET scan was performed ca. 60 min after tracer injection to assess metabolic activity in the brain, according to routine procedures at the Department of Nuclear Medicine of the University Hospital Zurich. Heart rate and blood pressure were recorded at baseline and throughout the procedure.

The procedure from the initial scan to the end of the final scan takes about 3.5 hours. Together with the 2 hours of preparation, participants spent about 5.5 hours on the study in total.

ELIGIBILITY:
Inclusion Criteria:

* Women and men that are between 50-75 years of age
* Post-menopausal status in women
* Normal body weight (BMI<30kg/m2)
* Non-smoker or not smoking since ≥ 5 years or occasional smokers.

Exclusion Criteria:

* Written informed consent was not provided
* History of arterial hypertension
* History of diabetes
* History of cardiovascular disease
* History of neurological disorders
* History of cancer (unless considered in remission since at least 5 years and not having necessitated a systemic chemotherapy and/or a brain radiotherapy)
* Use of steroids interfering with biomarker levels

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — We recruited healthy male and female volunteers, and gender identity was additionnally assessed using a gender score.
Study Population: We included healthy volunteers aged between 50-75 years old, post-menopausal in the case of women, recruited mainly in Switzerland.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-10-11 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Amygdala-to-cerebellum ratio of glycolytic metabolic activities (SUV/SUV) | 11-10-2021 to 20-11-2023
  Sex differences in the stress-related neural activity (SNA) assessed by 18F-FDG-PET and defined as the amygdala metabolic activity (AmygA, expressed as standard uptake value, SUV) corrected to the metabolic activity of the cerebellum (expressed as SUV), following the Trier Social Stress Test. The higher the AmygA/(cerebellum activity) ratio, the higher the SNA (no threshold for normality)
Difference between the rest and stress amygdala-to-cerebellum perfusion ratios (kBq/kBq) | 11-10-2021 to 20-11-2023
  Sex differences in the amygdala perfusion between rest and stress, assessed by 13N-NH3-PET and defined as the amygdala perfusion (AmygP, expressed as kiloBecquerel, kBq) corrected to the perfusion of the cerebellum (expressed as kBq), following the Montreal Imaging Stress Task. The higher the magnitude of the AmygP/(Cerebellum perfusion) modification at stress compared to rest, the higher the amygdala response to mental stress (no threshold for normality)
Myocardial flow reserve (MFR, no unit) | 11-10-2021 to 20-11-2023
  Sex differences in myocardial flow reserve (MFR) as determined by 13N-NH3-PET, during the Montreal Imaging Stress Task. MFR is defined as the ratio between MBF at stress and MBF at rest (no unit). The higher the MFR, the higher the myocardial perfusion modification during the stress task (no threshold).

SECONDARY OUTCOMES:
Amygdala-to-vmPFC ratio of glycolytic metabolic activities (SUV/SUV) | 11-10-2021 to 20-11-2023
  Sex differences in the stress-related neural activity (SNA) assessed by 18F-FDG-PET and defined as the amygdala metabolic activity (AmygA, expressed as standard uptake value, SUV) corrected to the metabolic activity of the ventromedial prefrontal cortex vmPFC (expressed as SUV), following the Trier Social Stress Test. The higher the AmygA/(vmPFC activity) ratio, the higher the SNA (no threshold for normality)
Difference between the rest and stress amygdala-to-vmPFC perfusion ratios (kBq/kBq) | 11-10-2021 to 20-11-2023
  Sex differences in the amygdala perfusion between rest and stress, assessed by 13N-NH3-PET and defined as the amygdala perfusion (AmygP, expressed as kiloBecquerel, kBq) corrected to the perfusion of the ventromedial prefrontal cortex (vmPFC, expressed as kBq), following the Montreal Imaging Stress Task. The higher the magnitude of the AmygP/(vmPFC perfusion) modification at stress compared to rest, the higher the amygdala response to mental stress (no threshold for normality)
Myocardial blood flow (MBF) at rest (mL/g/min) | 11-10-2021 to 20-11-2023
  Sex differences in myocardial blood flow (MBF, in mL/g/min) as determined by 13N-NH3-PET, during the control mode of the Montreal Imaging Stress Task. The higher the MBF, the higher the myocardial perfusion (no threshold).
Myocardial blood flow (MBF) at stress (mL/g/min) | 11-10-2021 to 20-11-2023
  Sex differences in myocardial blood flow (MBF, in mL/g/min) as determined by 13N-NH3-PET, during the stress mode of the Montreal Imaging Stress Task. The higher the MBF, the higher the myocardial perfusion (no threshold).
Heart-rate response (HRR, no unit) | 11-10-2021 to 20-11-2023
  Sex differences in the heart rate response (HRR), a surrogate for cardiac sympathetic activity, following each of the Montreal Imaging Stress Task and the Trier Social Stress Test. The HRR is defined as follows: HRR = ((Heart Rate at Stress) - (Heart Rate at Rest)/(Heart Rate at Rest)). The higher the HRR, the higher the cardiac sympathetic response to stress.
Salivary cortisol (mol/L) | 11-10-2021 to 20-11-2023
  Sex differences in the salivary cortisol response, a surrogate marker for the hypothalamic-pituitary-axis (HPA), to each of the Montreal Imaging Stress Task and the Trier Social Stress Test. The higher the cortisol increase, the higher the HPA response (no threshold).
Noradrenaline (mL/min) | 11-10-2021 to 20-11-2023
  Sex differences in the blood noradrenaline increase (mL/min) following the Trier Social Stress Task.
Adrenaline (mL/min) | 11-10-2021 to 20-11-2023
  Sex differences in the blood adrenaline increase (mL/min) following the Trier Social Stress Task.
Dopamine (mL/min) | 11-10-2021 to 20-11-2023
  Sex differences in the blood dopamine increase (mL/min) following the Trier Social Stress Task.
Spleen metabolic activity (SUV) | 11-10-2021 to 20-11-2023
  Sex differences in the spleen metabolic activity, a surrogate for systemic inflammation, following the Trier Social Stress Test, as assessed by 18F-FDG-PET, and expressed in standard uptake value (SUV). The higher the spleen SUV, the higher systemic inflammation.
Bone marrow metabolic activity (SUV) | 11-10-2021 to 20-11-2023
  Sex differences in the bone marrow metabolic activity, a surrogate for systemic inflammation, following the Trier Social Stress Test, as assessed by 18F-FDG-PET, and expressed in standard uptake value (SUV). The higher the bone marrow SUV, the higher systemic inflammation.
Aorta metabolic activity (SUV) | 11-10-2021 to 20-11-2023
  Sex differences in the thoracic aorta metabolic activity, a surrogate for aortic inflammation, following the Trier Social Stress Test, as assessed by 18F-FDG-PET, and expressed in standard uptake value (SUV). The higher the aorta SUV, the higher aorta inflammation.
Left ventricular ejection fraction (LVEF, %) | 11-10-2021 to 20-11-2023
  Sex differences in the left ventricular ejection fraction (LVEF, %) following the control and stress phases of the Montreal Imaging Stress Task.
C-reactive protein (CRP, mg/L) | 11-10-2021 to 20-11-2023
  Sex differences in C-reactive protein (CRP, in mg/L) collected at baseline and after the Trier Social Stress Test. The higher the CRP, the higher the inflammation.
Interleukin-2 (IL-2, pg/mL) | 11-10-2021 to 20-11-2023
  Sex differences in Interleukin-2 (IL-2), collected at baseline and after the Trier Social Stress Test. The higher the IL-2, the higher the inflammation.
Interleukin-4 (IL-4, pg/mL) | 11-10-2021 to 20-11-2023
  Sex differences in Interleukin-4 (IL-4) collected at baseline and after the Trier Social Stress Test. The higher the IL-4, the higher the inflammation.
Interleukin-6 (IL-6, pg/mL) | 11-10-2021 to 20-11-2023
  Sex differences in Interleukin-6 (IL-6) collected at baseline and after the Trier Social Stress Test. The higher the IL-6, the higher the inflammation.
Interleukin-8 (IL-8, pg/mL) | 11-10-2021 to 20-11-2023
  Sex differences in Interleukin-8 (IL-8) collected at baseline and after the Trier Social Stress Test. The higher the IL-8, the higher the inflammation.
Interleukin-10 (IL-10, pg/mL) | 11-10-2021 to 20-11-2023
  Sex differences in Interleukin-10 (IL-10) collected at baseline and after the Trier Social Stress Test. The higher the IL-10, the higher the inflammation.
Tumor necrosis factor (TNF, pg/mL) | 11-10-2021 to 20-11-2023
  Sex differences in Tumor necrosis factor (TNF, pg/mL) collected at baseline and after Trier Social Stress Test. The higher the TNF, the higher the inflammation.
Matrix metalloproteinase-9 (MMP9, pg/mL) | 11-10-2021 to 20-11-2023
  Sex differences in Matrix metalloproteinase-9 (MMP9, pg/mL), collected at baseline and after Trier Social Stress Test. The higher the MMP9, the higher the inflammation.
Monocyte Chemoattractant Protein-1 (MCP1, pg/mL) | 11-10-2021 to 20-11-2023
  Sex differences in Monocyte Chemoattractant Protein-1 (MCP1, pg/mL), collected at baseline and after Trier Social Stress Test. The higher the MCP1, the higher the inflammation.
Vascular Cell Adhesion Molecule (VCAM) | 11-10-2021 to 20-11-2023
  Sex differences in Monocyte Chemoattractant Protein-1 (MCP1, pg/mL), collected at baseline and after Trier Social Stress Test. The higher the VCAM, the higher the inflammation.
Gender score questionnaire | 11-10-2021 to 20-11-2023
  Sex differences in the self-perceived gender identity on a 0-to-100 scale, lower scores indicating a more pronounced "male gender" identity, higher scores indicating a more pronounced "female gender" identity. In addition to stratifying the analysis by sex, the role of gender on the results will be explored.

OTHER OUTCOMES:
Rate-Pressure-Product (RPP, in beats per minute x mmHg) | 11-10-2021 to 20-11-2023
  Sex differences in the rate-pressure-product (RPP, in beats per minute x mmHg) following the Montreal Imaging Stress Task, defined as the ratio between heart rate and systolic blood pressure. The higher the RPP, the higher the myocardial workload.
vmPFC-to-cerebellum ratio of glycolytic metabolic activities (SUV/SUV) | 11-10-2021 to 20-11-2023
  Sex differences in the metabolic activity of the ventromedial prefrontal cortex, assessed by 18F-FDG-PET, and defined as the vmPFC metabolic activity (expressed as standard uptake value, SUV) corrected to the metabolic activity of the cerebellum (expressed in SUV), following the Trier Social Stress Test. The higher the AmygA/(vmPFC activity) ratio, the higher the SNA (no threshold for normality)
Nail cortisol value (pg/mg) | 11-10-2021 to 20-11-2023
  Cortisol (pg/mg) as measured in the nails, a surrogate for chronic stress exposure.
General Anxiety Disorder (GAD-7) Questionnaire | 11-10-2021 to 20-11-2023
  Sex differences in the General Anxiety Disorder (GAD-7) questionnaire measuring anxiety severity on a 0-to-21 scale. The higher the score, the more pronounced anxiety symptoms.
Patient Health Questionnaire (PHQ-8) | 11-10-2021 to 20-11-2023
  Sex differences in the Patient Health Questionnaire (PHQ-8) assessing depressive symptoms on a 0-to-27 score. The higher the score, the more pronounced depressive symptoms.
Shortened Maastricht Exhaustion Questionnaire | 11-10-2021 to 20-11-2023
  Sex differences in the Shortened Maastricht Exhaustion Questionnaire assessing exhaustion levels on a 0-to-18 score. The higher the score, the more pronounced exhaustion symptoms.
Type D Personality (DS14) questionnaire | 11-10-2021 to 20-11-2023
  Sex differences in the Type D Personality (DS14) questionnaire on a 0-to-56 score. The higher the score, the more pronounced type D personality features.
Wagnild & Young Score resilience questionnaire | 11-10-2021 to 20-11-2023
  Sex differences in the Wagnild & Young Score resilience questionnaire on a 0-to-77 score. The higher the score, the more pronounced features of a resilient personality.
Perceived Stress Scale (PSS-4) questionnaire | 11-10-2021 to 20-11-2023
  Sex differences in the Perceived Stress Scale (PSS-4) questionnaire assessing stress levels in the previous months on a 0-to-16 scale. The higher the score, the higher the perceived stress.
Jenkins Sleep Scale (JSS-4) | 11-10-2021 to 20-11-2023
  Sex differences in the Jenkins Sleep Scale (JSS-4) evaluating sleep quality on a 0-to-16 scale.The higher the score the higher the sleep disturbances.
Trier Inventory for Chronic Stress (TICS) | 11-10-2021 to 20-11-2023
  Sex differences in the Trier Inventory for Chronic Stress (TICS) evaluating stress exposure in the preceding three months on a 0-to-228 scale. The higher the score, the more pronounced stress exposure.
Perceived stress | 11-10-2021 to 20-11-2023
  Sex differences in the perceived stress following each of the Montreal Imaging Stress Task and the Trier Social Stress Test, as self-assessed by the participants on a 0 to 7 Likert scale (0 indicating no perceived stress, and 7 indicating the highest possible stress perception).
Left ventricular stroke volume (LVSV, mL) | 11-10-2021 to 20-11-2023
  Sex differences in the left ventricular stroke volume (LVSV, mL), as measured by cardiac magnetic resonance, following the control and stress phases of the Montreal Imaging Stress Task.
Left ventricular end-systolic volume (LVESV, mL) | 11-10-2021 to 20-11-2023
  Sex differences in the left ventricular end-systolic volume (LVESV, mL), as measured by cardiac magnetic resonance, following the control and stress phases of the Montreal Imaging Stress Task.
Left ventricular end-diastolic volume (LVEDV, mL) | 11-10-2021 to 20-11-2023
  Sex differences in the left ventricular end-diastolic volume (LVEDV, mL), as measured by cardiac magnetic resonance, following the control and stress phases of the Montreal Imaging Stress Task.
Estradiol levels (pmol/L) | 11-10-2021 to 20-11-2023
  Estradiol levels (pmol/L) in blood collected at baseline.
Progesterone levels (nmol/L) | 11-10-2021 to 20-11-2023
  Progesterone levels (nmol/L) in blood collected at baseline.
Sex Hormone Binding Globulin (SHBG) levels (nmol/L) | 11-10-2021 to 20-11-2023
  Sex Hormone Binding Globulin (SHBG) levels (nmol/L) in blood collected at baseline.
Total testosterone levels (nmol/L) | 11-10-2021 to 20-11-2023
  Total testosterone levels (nmol/L) in blood collected at baseline.
Free testosterone levels (pmol/L) | 11-10-2021 to 20-11-2023
  Free testosterone levels (pmol/L) in blood collected at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Cathérine Gebhard, Professor, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided